CLINICAL TRIAL: NCT01172860
Title: Treatment of Inoperable Colorectal Cancer With Electrochemotherapy Through an Endoscopic System
Brief Title: Endoscopic Treatment of Inoperable Colorectal Cancer With the EndoVe System
Acronym: CCEE EndoVe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mercy University Hospital, Cork, Ireland (Other)
Collaborators: St. James's Hospital, Ireland (Other); The Adelaide and Meath Hospital (Other)
Responsible Party: Principal Investigator, Dr Declan Soden, Principal Investigator, Mercy University Hospital, Cork, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT:2012-001248-23
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer
Keywords: Inoperable; Colorectal; Endoscopic; Electroporation; Outpatient
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EndoVe treatment (Experimental): Use of the EndoVe device to safely and effectively ablate rectal tumor tissue
  Interventions: Device: EndoVe endoscopic electroporation

INTERVENTIONS:
Device: EndoVe endoscopic electroporation — The EndoVe device enables the endoscopic treatment of gastrointestinal tumor tissues. The device is placed on the tumor tissue and an electrical pulse of less than 1msec is delivered. The tumor tissue becomes permeabilised and absorbs much greater concentrations of the drug than the surrounding healthy tissue
  Other Names: EndoVe; Endoscope

SUMMARY:
A new approach to treating solid tumours (both operable and inoperable) has been carried out by the Cork Cancer Research Centre (CCRC) at the Mercy University Hospital, Cork, Ireland since 2002.

The approach simply allows a greater concentration of chemotherapy drugs to enter the tumour cells rather than healthy cells. The uptake of the chemotherapeutic drug directly by the tumour is aided through applying short electric pulses to the tumor mass (referred to as - Electrochemotherapy or ECT). The pulses make the tumour more porous which allows the drug easier access into the cancer cells, whereas other tissues and organs in the body remain relatively poor at absorbing the drug, thereby reducing the potential side effects on healthy tissues. This approach to date has been limited to skin based tumours due to the requirement for the electrodes to be placed directly in contact with the tumour. Procedures with electrochemotherapy have been applied to human patients in other countries of the EU, the US and Japan.

The drug concentration used is significantly reduced due to the more targeted absorption by the tumor and this significantly reduces side effects normally associated with chemotherapy.

A large number of preclinical and clinical Phase I and I/II studies have demonstrated the efficiency and safety of ECT. These studies have included patients with melanoma, head and neck squamous cell carcinoma, merkel cell carcinomas, basal cell carcinoma and adenocarcinoma nodules. Case reports concerning other primary tumours have also been reported.

The investigators have developed an endoscopic approach (EndoVe system) for delivering the electric pulses to internal cancers and are currently seeking to evaluate its efficacy in the treatment of inoperable colorectal cancer. The treatment procedure is similar to standard endoscopic colorectal examination (colonoscopy) with the added element of an intravenous injection of bleomycin followed after eight minutes by the delivery of electric pulses (each one less than 1msec in duration). The pulses are endoscopically delivered directly to the tumour mass. The entire procedure is minimally invasive and does not require intensive care follow up or stitches. If the treatment is successful the tumour will shrink in size in the weeks following the procedure.

The objective of this study is to investigate the efficacy and safety of this approach in reducing the size of the tumour.

DETAILED DESCRIPTION:
The objective is to conduct treatment in a minimally invasive manner (using the endoscope) and without the requirement for repeated doses of chemotherapy. The single dose of the drug used (15,000 IU/m2 x Body Surface Area of bleomycin) has been well tolerated in all patients treated previously with this approach to skin based cancers (in excess of 300 treatments since 2003 in our hospital). Therefore, it is anticipated that patients are unlikely to suffer side effects from the low concentration of drug used.

There are no known side effects of the instrument being tested. The pulse generator used has been certified by European electrical safety bodies charged with assessing compliance of new equipment with the present security rules for electrical devices. The electrical pulse generator has the CE mark and is approved for use clinically; the endoscopic electrodes used are a prototype system and are not currently CE approved.

The treatment is provided on an outpatient basis and does not involve an overnight stay. The procedure is very similar to a colonoscopy examination with the added element of a low dose chemotherapy drug being injected intravenously.

It reduces operative time; therefore there are fewer anaesthetic risks

At this time, the only option for patients with inoperable colorectal cancers is symptom relief e.g. a defunctioning colostomy or stent placement. Both carry a risk profile greater than the treatment with the EndoVe system.

Quicker recovery time- This is beneficial for the patient in terms of reduced exposure to the hospital environment through a shorter in-patient stay.

Research: The potential benefits of studying novel medical instruments in general include the development of new alternatives to conventional or existing therapies for certain cancers. In particular, the widespread availability of the novel instrument being tested here may lessen the requirement for more invasive procedures. It will reduce the amount of chemotherapy drug being used, therefore reducing the systemic effects as well as the side effects.

The approach is currently being applied to inoperable cases but in the future it may potentially be applied to both earlier stage cancers and other internal cancers e.g. oesophagus, stomach etc.

Because the treatment procedure is short (outpatient basis), it allows these patients greater time outside of the hospital environment to maximise and allowing for a greater quality of life (this for both individual patient and community at large).

If this treatment approach is proven to be safe and effective, patients with inoperable colorectal cancers will have a minimally invasive option for palliation of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified colorectal tumour.
2. Case reviewed by a multidisciplinary team (MDT) (surgery, radiology, oncology, gastroenterology) and there are no curable options with the standard of care. The MDT considers all available treatment options and enrolment to this study is agreed as being appropriate; Or the case is curable but patient refuses to undergo the standard of care. The MDT considers all possible alternatives, which are also discussed with the patient, and the MDT considers enrolment to this study as being the most appropriate option; Or patients with advanced local disease with impending obstruction on endoscopic evaluation who are otherwise not suitable for surgical intervention or stenting, the MDT would also consider these patients for enrolment into this study.
3. Men or women aged at least 18 years.
4. Performance status (Karnofsky > 60% or ECOG/WHO < 2).
5. Treatment free interval of at least 2 weeks after previously applied therapy.
6. Patients must be mentally capable of understanding the information given.
7. Patients must give written informed consent.
8. a) A female of Non-Childbearing potential (i.e. physiologically incapable of becoming pregnant) is eligible to participate in the study if she:

   * has had a hysterectomy
   * has had a bilateral oophorectomy (ovariectomy) - has had a bilateral tubal ligation
   * Is post-menopausal:

Exclusion Criteria:

1. Coagulation disorder
2. Patients with pre-existing renal dysfunction are excluded. [Note: Creatinine clearance will be measured for all patients. For Bleomycin treatment: creatinine clearance must be greater than 40ml/min.]
3. Patients with a clinically manifested arrhythmia or with a pacemaker
4. Patients with epilepsy.
5. Pregnancy or lactation/breastfeeding.
6. Patient known to be Hepatitis B/C or HIV positive.
7. Concurrent treatment with an investigational medicinal product or participation in another clinical study.
8. Patients who have undergone a regime of Bevacizumab in the previous 4 weeks.
9. Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.
10. Highly inflamed colon tissue which is ulcerated and bleeding.

    Additional exclusion criteria specifically regarding patients where Bleomycin is study drug:
11. Contraindications for bleomycin use including acute pulmonary infection and severe pulmonary disease.
12. Contraindication for bleomycin use: allergic reactions to bleomycin observed in previous treatment.
13. Contraindication for bleomycin use: if cumulative dose of 250mg BLM/m2 was previously exceeded.

    Additional exclusion criteria specifically regarding patients where Cisplatin is study drug:
14. Patients with hypersensitivity to Cisplatin or other platinum compounds or to any of the excipients are to be excluded from receiving Cisplatin for the study.
15. Cisplatin is contraindicated in combination with live vaccines, including yellow fever vaccine.
16. Cisplatin is contraindicated in combination with phenytoin in prophylactic use.
17. Cisplatin is contraindicated in patients with myelosuppression.
18. Cisplatin is contraindicated in patients in a dehydrated condition (pre- and post-hydration is required to prevent serious renal dysfunction).
19. Cisplatin is contraindicated in patients with a pre-existing hearing impairment.
20. Cisplatin is contraindicated in patients with neuropathy caused by cisplatin.
21. Contraindication for Cisplatin use: Allergic reactions to Cisplatin observed in previous treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Tumor regression | 3 months
  Follow up examination of tumor volume following treatment via endoscopy and transrectal ultrasound.
treatment safety | 3 months
  Evaluate safety of treatment approach at regular checkup intervals following treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy University Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gargiulo M, Moio M, Monda G, Parascandolo S, Cubicciotti G. Electrochemotherapy: actual considerations and clinical experience in head and neck cancers. Ann Surg. 2010 Apr;251(4):773. doi: 10.1097/SLA.0b013e3181d64b81. No abstract available. PMID 20375711
- [Background] Moller MG, Salwa S, Soden DM, O'Sullivan GC. Electrochemotherapy as an adjunct or alternative to other treatments for unresectable or in-transit melanoma. Expert Rev Anticancer Ther. 2009 Nov;9(11):1611-30. doi: 10.1586/era.09.129. PMID 19895245
- [Background] Campana LG, Mocellin S, Basso M, Puccetti O, De Salvo GL, Chiarion-Sileni V, Vecchiato A, Corti L, Rossi CR, Nitti D. Bleomycin-based electrochemotherapy: clinical outcome from a single institution's experience with 52 patients. Ann Surg Oncol. 2009 Jan;16(1):191-9. doi: 10.1245/s10434-008-0204-8. Epub 2008 Nov 6. PMID 18987914
- [Background] Quaglino P, Mortera C, Osella-Abate S, Barberis M, Illengo M, Rissone M, Savoia P, Bernengo MG. Electrochemotherapy with intravenous bleomycin in the local treatment of skin melanoma metastases. Ann Surg Oncol. 2008 Aug;15(8):2215-22. doi: 10.1245/s10434-008-9976-0. Epub 2008 May 23. PMID 18498012
- [Background] Sadadcharam M, Soden DM, O'sullivan GC. Electrochemotherapy: an emerging cancer treatment. Int J Hyperthermia. 2008 May;24(3):263-73. doi: 10.1080/02656730701832334. PMID 18393004
- [Background] Larkin JO, Collins CG, Aarons S, Tangney M, Whelan M, O'Reily S, Breathnach O, Soden DM, O'Sullivan GC. Electrochemotherapy: aspects of preclinical development and early clinical experience. Ann Surg. 2007 Mar;245(3):469-79. doi: 10.1097/01.sla.0000250419.36053.33. PMID 17435555
- [Background] Mir LM, Morsli N, Garbay JR, Billard V, Robert C, Marty M. Electrochemotherapy: a new treatment of solid tumors. J Exp Clin Cancer Res. 2003 Dec;22(4 Suppl):145-8. PMID 16767921
- [Background] Byrne CM, Thompson JF. Role of electrochemotherapy in the treatment of metastatic melanoma and other metastatic and primary skin tumors. Expert Rev Anticancer Ther. 2006 May;6(5):671-8. doi: 10.1586/14737140.6.5.671. PMID 16759159
- [Background] Soden DM, Larkin JO, Collins CG, Tangney M, Aarons S, Piggott J, Morrissey A, Dunne C, O'Sullivan GC. Successful application of targeted electrochemotherapy using novel flexible electrodes and low dose bleomycin to solid tumours. Cancer Lett. 2006 Feb 8;232(2):300-10. doi: 10.1016/j.canlet.2005.03.057. Epub 2005 Jun 16. PMID 15964138
- [Background] Snoj M, Rudolf Z, Cemazar M, Jancar B, Sersa G. Successful sphincter-saving treatment of anorectal malignant melanoma with electrochemotherapy, local excision and adjuvant brachytherapy. Anticancer Drugs. 2005 Mar;16(3):345-8. doi: 10.1097/00001813-200503000-00015. PMID 15711188